CLINICAL TRIAL: NCT06645301
Title: Exploratory Clinical Study Initiated by Researchers on the Safety and Preliminary Efficacy of BGT007 in Treating Patients with Recurrent/refractory Gastrointestinal Malignancies
Brief Title: BGT007 Treatment for Recurrent/refractory Gastrointestinal Malignancies
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: BioSyngen Pte Ltd (Industry)
Collaborators: South China Hospital of Shenzhen University (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BR-BGT007-001
Record Dates: First submitted 2024-10-15; First posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Colorectal Cancer; Pancreatic Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- BGT007 (Experimental): Intravenous infusion
  Interventions: Biological: Group A; Biological: Group B

INTERVENTIONS:
Biological: Group A — BGT007 3.0×10^8cells,Intravenous infusion，3 subject is planned to be enrolled
Biological: Group B — BGT007 6.0×10^8cells,Intravenous infusion，6 subject is planned to be enrolled

SUMMARY:
This study is an exploratory research on single arm, open, and improved "3+3" dose escalation. BGT007 will explore two dose groups, namely (Group A: 3.0X10 ^ 8 3 cases, Group B: 6.0X10 ^ 8 3 cases), and receive the same dose infusion after observing lower adverse reactions and initial benefits (SD or PR), with an interval of one month. Each subject can receive a maximum of 3 infusions in total.

DETAILED DESCRIPTION:
Main research objectives:

Evaluate the safety and tolerability of BGT007 in treating patients with recurrent/refractory multiple gastrointestinal malignancies;

Secondary research objective:

1. Evaluate the pharmacokinetic (PK) characteristics of BGT007;
2. Evaluate the preliminary effectiveness of BGT007 product.

ELIGIBILITY:
Inclusion Criteria:

* 1: Voluntarily sign a written informed consent form;
* 2: Age ≥ 18 years old and ≤ 75 years old, both male and female are acceptable;
* 3: Expected survival period ≥ 3 months;
* 4: The physical fitness score of the Eastern Cooperative Oncology Group (ECOG) is 0 or 1;
* 5: Biopsy specimens or pathological paraffin sections (within 3 years prior to signing the informed consent form): target tests are both positive;
* 6: According to the RECIST v1.1 solid tumor evaluation criteria, there must be at least one measurable lesion, and the longest diameter evaluated by CT or MRI imaging in the baseline period must be ≥ 10 mm (excluding lymph nodes, whose short diameter must be ≥ 15 mm);
* 7: Advanced pancreatic cancer or colorectal cancer confirmed by histology or cytology, which has progressed through second-line or above standard treatment, or is intolerant of standard treatment, or has no standard treatment; Definition of intolerance: According to CTCAE V5.0, during the treatment process, there is a hematological toxicity of ≥ Grade IV, non hematological toxicity of ≥ Grade III, or damage to major organs such as the heart, liver, and kidneys of ≥ Grade II; The definition of treatment failure: disease progression (PD) during the treatment process or recurrence after treatment (including postoperative recurrence);
* 8: Can establish a single or intravenous blood collection pathway, and there are no other contraindications for blood cell isolation;
* 9: Having sufficient organ and bone marrow functions
* 10: Medical contraceptive measures. Female subjects of childbearing age must undergo a pregnancy test within 72 hours before the first administration, and the result must be negative.

Exclusion Criteria:

* 1: Active central nervous system metastases (excluding those that have been treated and stabilized);
* 2: HIV positive, HBsAg positive with HBV DNA copy number positive (greater than the detection limit), HCV antibody positive and HCV RNA positive, syphilis non-specific antibody (RPR or TRUST) positive;
* 3: Individuals with mental or psychological disorders who are unable to cooperate with treatment and efficacy evaluation;
* 4: Subjects with severe autoimmune diseases and long-term use of immunosuppressants;
* 5: Within the 14 days prior to enrollment, there were active or uncontrollable infections that required systemic treatment;
* 6: Any unstable systemic disease (including but not limited to): active infection (excluding local infection); Unstable angina pectoris; Cerebrovascular ischemia or cerebrovascular accident (within 6 months prior to screening); Myocardial infarction (within 6 months prior to screening); Congestive heart failure (NYHA classification ≥ III); Severe arrhythmia requiring medication treatment; Heart disease requiring treatment or uncontrolled hypertension after treatment (blood pressure>160mmHg/100 mmHg);
* 7: Functional impairment of important organs such as lungs, brain, and kidneys;
* 8: The subjects have undergone major surgery or severe trauma within 4 weeks prior to receiving treatment with the investigational product, or are expected to undergo major surgery during the study period;
* 9: Received any systemic chemotherapy, immunotherapy, or small molecule targeted therapy within 2 weeks prior to single collection or within 5 half lives (whichever is shorter);
* 10: Received treatment with chimeric antigen receptor modified T cells (including CAR-T and TCR-T) within six months;
* 11: Severe allergies or a history of allergies;
* 12: Subjects requiring anticoagulant therapy;
* 13: Pregnant or lactating women, or those with a pregnancy plan within six months (for both men and women)
* 14: Researchers believe that there are other reasons why treatment providers cannot be included.

Ages: 17 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-11-30 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Dose-Limiting Toxicity (DLT) | From the infusion (Day 0) to Day 28
  DLT is defined as the following adverse events related to the investigational drug(definitely related, likely related,possibly related) that occur within 28 days after administration of BGT007 (using CTCAE 5.0 or CRS grading criteria): (1) hematological toxicity; (2) Grade 3 non hematological toxicity lasting for more than 7 days, or ≥ Grade 4 non hematological toxicity, regardless of duration, but excluding the following situations; (3)Cytokine Release Syndrome(CRS)
Maximum Tolerated Dose(MTD) | From the infusion (Day 0) to Day 28
  The highest dose of DLT observed in subjects with less than 2/6 (at least 6 subjects in this experimental group received BGT007 administration and completed DLT observation)

CONTACTS AND LOCATIONS:
Overall Officials: Mingyong Han, PhD, Principal Investigator — South China Hospital of Shenzhen Univercity; Yuqing Li, PhD, Principal Investigator — South China Hospital of Shenzhen Univercity